CLINICAL TRIAL: NCT02212171
Title: TRIAP: Is Triage by Healthcare Mini-teams Effective to Improve Efficiency in Primary Health Care?
Acronym: TRIAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Roberto Gonzalez Santisteban, Physician, Basque Health Service
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TRIAP; 2011111131 (Other Grant/Funding Number: Basque Health Goverment)
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Organization of Health Service
MeSH Terms: interventions — Malononitrile dimer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TRIAP intervention (Experimental)
  Interventions: Other: TRIAP
- Usual care (No Intervention): Usual care: Patients in the control group will be treated according to Osakidetza recommendations.

INTERVENTIONS:
Other: TRIAP — The primary healthcare professionals organised in healthcare mini-teams, composed of 2 doctors, 2 nurses and 1 member of the administrative staff.
  1. Administrative staff:
     Following a flow chart, they will refer patients with mild self-limiting illnesses as well as consultations regarding chronic disorders in adults to the nurses. They will also perform administrative tasks such as the printing of prescriptions, sick leave reports and medical notes (justifying absence), etc.
  2. Nursing staff:
     They will carry out activities focused on health promotion, self-management and de-medicalisation during visits from patients with mild self-limiting illnesses as well as appointments for chronic diseases in adults.
  3. GP:
  They will develop the new portfolio of services: health promotion, joint review of patient medical records by doctors and nurses to improve the management of certain groups of patients, and organization of minor surgery services, etc.
  Arms: TRIAP intervention

SUMMARY:
Background: With new challenges for healthcare, there is a clear consensus among experts on the need to introduce changes in the organization of care in health centres to address the problems of over-attendance, bureaucratization and other emerging issues that require growing amounts of attention. However, there has been insufficient research into possible models and the impact of their adoption.

The objective is to assess the feasibility and effectiveness of the TRIAP intervention, a new organizational model based on triage and healthcare mini-teams (two general practitioners/pediatricians, two nurses and one member of the administrative staff) compared to the current model, aiming to achieve a correct classification of the healthcare needs of the primary care population and direct them to the most suitable professional.

In addition, the implementation research objective is to identify the facilitators for and barriers to the implementation of the intervention in the context of primary care.

Methods/ design: This is a quasi-experimental controlled clinical trial to be performed in 14 healthcare mini-teams (7 intervention and 7 control groups) from 8 health centres in the Basque Healthcare Service (Osakidetza) Interior Health Region.

The results will be assessed using the data on morbidity-adjusted attendance of users to their family doctor, number of referral, addition of new activities to the portfolio of services, and patient perception and professional satisfaction. All the variables will be measured at baseline and at the end of the intervention, 24 months later.

Using covariance analysis models, the investigators will estimate the effect attributable to the intervention by analyzing differences in changes between the two groups, and calculating the 95% confidence interval, adjusting the comparisons for baseline values. The investigators will also adjust for potential confounding and effect-modifying variables.

Nominal groups will be held at the end of the intervention with the participation of all the agents involved in intervention centres to identify the facilitators for and barriers to the implementation of the intervention.

Discussion: There is a need to develop new forms of organization in primary care services to respond to new healthcare demands. To pursue this aim, changes have to be introduced in the organization of healthcare within health centres, redefining the roles of primary care professionals and refocusing their activity towards population health needs, seeking greater efficiency in health services.

ELIGIBILITY:
Inclusion Criteria:

* The study populations are patients of the seven mini-teams established, these professionals being responsible for the GP lists in the health centres of San Miguel in Basauri, Miraballes and Ondarroa, and the paediatric list in Etxebarri health centre. The control units are from the health centres of Basauri-Ariz, Arratia, Amorebieta and Bermeo, all located in the Interior Health Region.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Actual)
Dates: Start 2012-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Patients attendance | Baseline and at 24 months
  Number of visits of the patients to their GP and paediatricians in accordance to the Adjusted Clinical Groups [ACG] Case-Mix System.
  The patients will be classified using the ACG system, on the basis of their age, sex and ICD-9-CM codes of health problems diagnosed over a year in visits to their GP/paediatrician. The ACG case-mix system was designed by researchers at Johns Hopkins University, originally for care on an outpatient basis, and classifies the population into around 100 self-excluding categories.
  Regardless of the number of contacts with the healthcare services, each person is classified every year into a single ACG depending on their age, sex, and combination of diagnoses they were assigned over the previous 12 months. For this study, we will use the ACG Assignment Software version 7.00.
  All the tasks performed will be recorded in the Osabide computer system of the Basque Health Service.

SECONDARY OUTCOMES:
Patients referral: number of patient referrals by GPs and paediatricians in accordance to the Adjusted Clinical Groups [ACG] Case-Mix System. | Baseline and at 24 months
New activities added to the current portfolio of services | Baseline and at 24 months
  Number of programmed activities of health promotion, joint review of medical records by the doctors and nurses to improve the management of certain groups of patients, minor surgery services in PC, activities for achieving a comprehensive approach to managing non-surgical osteomuscular disorders and the use of ultrasound scans.
Patient satisfaction | Baseline and at 24 months
  Measured using the Primary Care Assessment Tool (PCAT) Pasarín MI et al. Evaluation of primary care: The "Primary Care Assessment Tools - Facility version" for the Spanish health system. Gac Sanit. 2013 Jan-Feb;27(1):12-8.
Satisfaction of health professionals | Baseline and at 24 months
  In terms of professional quality of life measured using the Professional Quality of Life questionnaire (PQL-35).
  Cabezas, C. La calidad de vida de los profesionales. FMC. 2000;7 (Supl 7):53-68.

CONTACTS AND LOCATIONS:
Locations (1):
- Basque Healthcare Service, Vitoria-Gasteiz, Spain